CLINICAL TRIAL: NCT00068289
Title: A Phase II Trial of PS-341 (NSC-681239) in Patients With Platinum-Treated Extensive Stage Small Cell Lung Cancer
Brief Title: Bortezomib in Treating Patients With Recurrent or Refractory Extensive-Stage Small Cell Lung Cancer Previously Treated With Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000320527; SWOG-S0327
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have recurrent or refractory extensive-stage small cell lung cancer that was previously treated with platinum-based chemotherapy (such as cisplatin, carboplatin, or oxaliplatin).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of bortezomib, in terms of response rate (confirmed and unconfirmed, complete and partial), in patients with recurrent or refractory extensive stage small cell lung cancer previously treated with platinum-based therapy.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the overall survival of patients treated with this drug.
* Correlate selected molecular markers with outcomes in patients treated with this drug.

OUTLINE: Patients are stratified according to platinum-sensitivity status (platinum sensitive [temporarily closed to accrual as of 8/1/04] vs platinum refractory [temporarily closed to accrual as of 6/1/04]).

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 40-80 patients (20-40 per stratum) will be accrued for this study within 0.5-1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung cancer

  * Diagnosis by sputum cytology allowed provided it is confirmed by an independent pathologic review
  * Clinical evidence of recurrent or refractory disease does not require a confirmatory biopsy
* Measurable disease by plain radiographs, CT scan, or MRI

  * Prior radiotherapy to measurable disease allowed provided there is evidence of disease progression by CT scan OR there is measurable disease outside of the radiotherapy field
* Must have received a prior platinum-based chemotherapy regimen and meet criteria for 1 of the following:

  * Platinum-sensitive disease, defined as an initial response with subsequent progression more than 90 days after last platinum treatment (temporarily closed to accrual as of 8/1/04)
  * Platinum-refractory disease, defined as no response to or progression during platinum treatment or subsequent progression no more than 90 days after last platinum treatment (temporarily closed to accrual as of 6/1/04)
* Brain and/or leptomeningeal metastases are allowed provided all of the following are true:

  * Asymptomatic on neurological exam
  * No concurrent corticosteroids for symptom control
  * No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin or phenobarbital)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine no greater than upper limit of normal OR
* Creatinine clearance at least 60 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No symptomatic sensory neuropathy greater than grade 1
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any other adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy to measurable lesions

Surgery

* At least 14 days since prior thoracic or other major surgery and recovered

  * Must have disease outside of the prior surgical resection area OR new lesion must be present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD — University of California, Davis; Angela Davies, MD — University of California, Davis
Locations (91):
- United States (90):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Salisbury, Salisbury, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lara PN Jr, Chansky K, Davies AM, Franklin WA, Gumerlock PH, Guaglianone PP, Atkins JN, Farneth N, Mack PC, Crowley JJ, Gandara DR. Bortezomib (PS-341) in relapsed or refractory extensive stage small cell lung cancer: a Southwest Oncology Group phase II trial (S0327). J Thorac Oncol. 2006 Nov;1(9):996-1001. PMID 17409985
- [Result] Johl J, Chansky K, Lara PN, et al.: The proteasome inhibitor PS-341 (bortezomib) in platinum (plat)-treated extensive-stage small cell lung cancer (E-SCLC): a SWOG (0327) phase II trial. [Abstract] J Clin Oncol 23 (Suppl 16): A-7047, 632s, 2005.
- [Derived] Lara PN Jr, Moon J, Redman MW, Semrad TJ, Kelly K, Allen JW, Gitlitz BJ, Mack PC, Gandara DR. Relevance of platinum-sensitivity status in relapsed/refractory extensive-stage small-cell lung cancer in the modern era: a patient-level analysis of southwest oncology group trials. J Thorac Oncol. 2015 Jan;10(1):110-5. doi: 10.1097/JTO.0000000000000385. PMID 25490004